CLINICAL TRIAL: NCT03043183
Title: The Effect of Perioperative Nutritional Status on Enhanced Recovery After Surgery for Gastric Cancer
Brief Title: Enhanced Recovery After Surgery(ERAS) for Gastric Cancer and Perioperative Nutritional Status
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Quan Wang, Director, The First Hospital of Jilin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ERAS AND Nutritional Status
Record Dates: First submitted 2017-02-02; First posted 2017-02-03 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Nutrition Disorders
Keywords: gastric cancer; Enhanced recovery after surgery
MeSH Terms: conditions — Nutrition Disorders; Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperational nutrition support group (Experimental): Scored patient-generated subjective global assessment(PG-SGA) ≥2，<9 Oral enteral nutrition support（25 kcal/kg or 1.5 g protein/kg） for 3 days before operation
  Interventions: Procedure: perioperational nutrition surpport
- Conventional group (No Intervention): PG-SGA ≥2，<9

INTERVENTIONS:
Procedure: perioperational nutrition surpport — Oral enteral nutrition support（25 kcal/kg or 1.5 g protein/kg） for 3 days before operation
  Arms: Preoperational nutrition support group

SUMMARY:
This study is a prospective, single-center, randomized controlled trial. The study protocol was approved by the Ethics Committee at the First Hospital of Jilin University.The perioperation nutritional status will be assessed in gastric cancer patients within ERAS protocols.The ERAS patients were randomly divided into perioperational nutrition support group and conventional pathway group . Inter-group differences were evaluated for nutritional index,clinical recovery index, complications etc.

ELIGIBILITY:
Inclusion Criteria:

* A preoperative cancer stage of T2, T3, T4, Any N, M0 without digestive obstruction confirmed by whole body CT scan, which could be treated with laparoscopic gastrectomy;
* age 18-75 years;
* pathologic confirmation of gastric adenocarcinoma by endoscopic biopsy;
* normal hematological, renal, hepatic, and cardiac parameters,American Society of Anesthesiology (ASA) score < III without severe systemic disease;
* no history of treatment with neoadjuvant chemotherapy and/or radiotherapy
* PG-SGA score ≥2，<9

Exclusion Criteria:

* patients requiring conversion to open gastrectomy
* excessive bleeding (˃ 500 mL);and patients opting out of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2017-03-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
complication | 30 days after operation
  fever；wound infection；post-operation bleeding；ileus；stenosis；leakage